CLINICAL TRIAL: NCT03766789
Title: Use of a Smartphone Digital Application as a Tool to Increase Adherence to Medical Treatment in Patients Who Underwent Hospitalization for Acute Coronary Syndrome.
Brief Title: Use of a Smartphone Application to Increase Adherence to Medical Treatment in Patients With an Acute Coronary Syndrome.
Acronym: ADHERENCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Cardiovascular de Buenos Aires (Other)
Responsible Party: Principal Investigator, Juan Pablo Costabel, Principal Investigator., Instituto Cardiovascular de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: A0001
Record Dates: First submitted 2018-12-02; First posted 2018-12-06 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Adherence, Medication
Keywords: Adherence, Medication, Therapy
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): They will receive the cell phone application, as reminder of medications time and dose.
  Interventions: Device: Cell phone application
- Control (No Intervention): Patients will receive standard of care recommendations.

INTERVENTIONS:
Device: Cell phone application — cell phone to organize medications
  Arms: Intervention

SUMMARY:
ADHERENCE is a randomized unicentric study that will be carried out from a monovalent center of cardiology of the Autonomous City of Buenos Aires. Patients will be randomized hospitalization for acute coronary syndromes (ACS) with and without ST segment elevation at the time of hospital discharge to receive access to a digital application for smartphones or receive written instructions regarding the taking of medication as prescribed by doctors . They will have a total follow-up period of 90 days, in which the adherence to medical treatment will be evaluated through a questionnaire validated for that purpose.

The objective of the study is to demonstrate that the use of a digital platform for smartphones increases the adherence to medical treatment by 30% in relation to the group without intervention

DETAILED DESCRIPTION:
The World Health Organization (WHO) states that poor adherence to long-term medical treatments severely compromises their effectiveness, with an expected adherence of 50% in developed countries and less in developing countries. This non-compliance to medical treatment tends to increase as the global burden of chronic diseases increases, where not only the rational use of medicines but also compliance with prescribed treatments becomes vitally important. So it is of interest to highlight the importance not only of the clarity of the medical prescription at the time of hospital discharge but of compliance with it in the out-of-hospital setting.

The lack of adherence to medical treatment is a difficult problem to solve, and this could partially explain the ineffectiveness of the treatments administered by the health system. Adherence is greater in the acute phase of the disease2, presenting a marked decrease within 3 to 6 months of treatment3. In order to avoid this problem, multiple interventions have been studied without evidence of significant benefits or clinical impact.

The "Medication Reminder" application will be used as a digital tool for smartphones, which is available for different commercial software platforms, free download. The intervention group will have the installation of the aforementioned platform on your smartphone, loading the list of your medication, as well as an alarm in the hours proposed for the shot. When the warning is presented, the patient will have a warning by which he will have to accept or reject the taking of the medication; to reject it, the reminder will remain present for 24hs and then it will be automatically deleted. At the end of the day, the patient can access an analysis of daily compliance and thus perform a self-monitoring. The control group will receive the standard of care, consisted of a written list of medications.

We will evaluate the adherence to medications at 3 months as primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Acquire hospitalization for acute coronary syndromes (ACS) with and without ST segment elevation.
* Have access to a smartphone in order to access the digital application provided.
* Have the possibility to follow up after 90 days.
* Sign the informed consent administered in writing prior to inclusion in the clinical trial.

Exclusion Criteria:

* Patients with coronary lesions with a revascularization planned (revascularization in stages).
* Severe limitation of mobility (amputation, degenerative myopathies, musculoskeletal disorders).
* Total or intermediate dependency for carrying out tasks of daily life according to the validated Katz questionnaire of Activities of Daily Life (ADL). -

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2019-01-27 (Estimated)

PRIMARY OUTCOMES:
Adherence to treatment | 3 months
  Rate of patients in each arm with adherence to medical treatment defined by the Morisky Green scale.
  The eight-item Morisky Medication Adherence Scale (MMAS-8) is a structured self-report measure of medication-taking behavior that has been widely used in various cultures. The first seven items are dichotomous response categories with yes or no and the last item was a five point Likert response. The adherence to medications is higher in patients with higher scale values (values from 0 to 8). A patient is consider to have good adherence when score is perfect (8 points)

SECONDARY OUTCOMES:
Impact in clinical events | 3 months
  Rate of patients in each arm with the combined event of re-hospitalizations for acute coronary syndromes, consultations to the medical emergency system or not planned visits to clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Costabel, MD, Principal Investigator — Chief of coronary care unit
Locations (1):
- Juan Pablo Costabel, Buenos Aires, Argentina